CLINICAL TRIAL: NCT00769184
Title: A Steroid-Sparing Effect of Supplemental LCD Treatment in Patients With Moderate-to-Severe Localized Psoriasis Lesions: a Pilot Study.
Brief Title: Combining Topical Corticosteroid and LCD Treatment for Localized Plaque Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeoStrata Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-LCDSTRD
Record Dates: First submitted 2008-10-07; First posted 2008-10-09 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-07

CONDITIONS: Psoriasis
Keywords: chronic plaque psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adrenal Cortex Hormones; Clobetasol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corticosteroid + LCD (Experimental): corticosteroid and LCD treatment (2 weeks), LCD alone treatment (4 weeks)
  Interventions: Drug: Corticosteroid; Drug: LCD
- Corticosteroid + Placebo (Placebo Comparator): corticosteroid and placebo treatment (2 weeks), placebo alone treatment (4 weeks)
  Interventions: Drug: Corticosteroid; Other: Placebo

INTERVENTIONS:
Drug: Corticosteroid — One side of body:
  clobetasol: 2 applications / day along with LCD application 2 applications/day
  Other Names: clobetasol
Other: Placebo — One side of body:
  Placebo Solution: 2 applications / day along with clobetasol 2 applications/day
  Arms: Corticosteroid + Placebo
Drug: LCD — One side of body:
  LCD Solution: 2 applications / day along with clobetasol 2 applications/day
  Other Names: liquor carbonis distillate
  Arms: Corticosteroid + LCD

SUMMARY:
This is a 12 week bilateral study, consisting of 6 weeks of treatment and 6 weeks of follow-up. The purpose of the study is to compare the safety and effectiveness of combining and then following a high potency topical corticosteroid treatment with LCD treatment for moderate-to-severe localized plaque psoriasis.

DETAILED DESCRIPTION:
Superpotent topical corticosteroids such as clobetasol propionate are highly effective in treating plaque psoriasis but are not indicated for long term use due to their side effects. Therefore, steroid-sparing combination and sequential regimens, in which the corticosteroid gets supplemented with a non-steroid medication, such as calcipotriol or tazarotene, have become the standard of care, especially in the management of localized psoriasis lesions. A new steroid-free 15% liquor carbonis distillate (LCD) solution (Psorent) was recently found to be more successful than 0.005% calcipotriol cream (Dovonex) at improving and delaying worsening of psoriasis symptoms in a controlled clinical trial. The goal of this pilot study is to evaluate if this LCD solution can be used in combination with acute topical corticosteroid therapy as a new steroid-sparing / enhancing regimen. We hope to explore the compatibility, patient tolerability, and clinical benefit of using LCD solution during and after treatment with clobetasol propionate in adults with moderate to severe plaque psoriasis. This is a randomized, double-blind, vehicle-controlled, bilateral study. Men and women 18 years of age or older, with chronic plaque psoriasis affecting less than or equal to 10% body surface area (BSA) in areas other than the scalp, face, palms, soles, axillae, and groin, are recruited. Those with a Physician Global Assessment (PGA) score greater than 3 and are in general good health will qualify as candidates. On one side of the body, LCD solution and clobetasol propionate will be administered twice daily for the first 2 weeks of treatment, followed by 4 weeks of LCD solution only, followed by 6 weeks of no treatment. On the second half of the body, subject will apply a vehicle solution and clobetasol propionate twice daily for the first 2 weeks, only the vehicle solution twice daily for the next four weeks, and then no treatment for the next 6 weeks. Subjects will be evaluated at weeks 2, 4, 6, 8, 10 and 12. investigators will use the PGA scale [Clear (0) - Severe (5)] to determine treatment effects as well as Target Lesion assessments of Erythema, Scaling, Induration and overall severity [None (0) - Very Severe (4)]. patients will also be required to complete Self-Assessment questionnaires on their psoriasis [None (0) - Severe (6)]. as well as an assessment of the study solution [Excellent (9) - Poor (1)]. . Photographs will be taken at each study visit and adverse events will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* able to provide written informed consent
* able to attend study visits, apply medications, and follow instructions
* moderate to severe localized plaque psoriasis lesions (<10% BSA on each side of the body)

Exclusion Criteria:

* other current treatments for psoriasis
* hypersensitivity to steroids, liquor carbonis detergens, alcohol, fragrance
* pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Bagel, MD, Principal Investigator — Psoriasis Treatment Center of Central New Jersey
Locations (1):
- Windsor Dermatology, East Windsor, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Corticosteroid + LCD (Left), Corticosteroid + Placebo (Right): Corticosteroid + LCD on left side of body, Corticosteroid + Placebo on right side of body (n=7).
  On left side: Corticosteroid + liquor carbonis distillate (LCD) treatment applied, twice a day, for 2 weeks, then LCD-only, twice a day, for 4 weeks, then no treatment for 6 weeks
  On right side: Corticosteroid and placebo vehicle solution, twice a day, for 2 weeks, then placebo vehicle solution-only, twice a day, for 4 weeks, then no treatment for 6 weeks
- Corticosteroid + LCD (Right), Corticosteroid + Placebo (Left): Corticosteroid + LCD on right side of body, Corticosteroid + Placebo on left side of body (n=8).
  On right side: Corticosteroid + liquor carbonis distillate (LCD) treatment applied, twice a day, for 2 weeks, then LCD-only, twice a day, for 4 weeks, then no treatment for 6 weeks
  On left side: Corticosteroid and placebo vehicle solution, twice a day, for 2 weeks, then placebo vehicle solution-only, twice a day, for 4 weeks, then no treatment for 6 weeks
Period: Corticosteroid + LCD/ +Placebo (2 Weeks)
Arm/Group | Corticosteroid + LCD (Left), Corticosteroid + Placebo (Right) | Corticosteroid + LCD (Right), Corticosteroid + Placebo (Left)
Started | 7 | 8
Completed | 6 | 7
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: +LCD / +Placebo Only (4 Weeks)
Arm/Group | Corticosteroid + LCD (Left), Corticosteroid + Placebo (Right) | Corticosteroid + LCD (Right), Corticosteroid + Placebo (Left)
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0
Period: No Treatment (6 Weeks)
Arm/Group | Corticosteroid + LCD (Left), Corticosteroid + Placebo (Right) | Corticosteroid + LCD (Right), Corticosteroid + Placebo (Left)
Started | 6 | 7
Completed | 5 | 6
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Fifteen patients with localized chronic plaque psoriasis (less than or equal to 6% BSA and PGA score greater than or equal to 3) were enrolled. Eleven patients completed the study. Three patients were removed due to an adverse event, and 1 patient was lost to follow-up after week 2.
Groups:
- Corticosteroid+LCD vs Corticosteroid+Placebo: one side of body: corticosteroid and liquor carbonis distillate (LCD) treatment applied twice a day, for 2 weeks, then LCD-only twice a day, for 4 weeks, then no treatment for 6 weeks
  opposite side of body: corticosteroid and placebo vehicle solution twice a day, for 2 weeks, then placebo vehicle solution-only twice a day, for 4 weeks, then no treatment for 6 weeks
Arm/Group | Corticosteroid+LCD vs Corticosteroid+Placebo
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Are Clear (PGA Score 0) or Have Minimal Disease (PGA Score 1) on Each Treated Side at Each Visit.
Description: Those patients that have reached a PGA score of zero [PGA scale: clear (0) - very severe (5)], and are considered clear of chronic plaque psoriasis, or have reached a PGA score of 1, with minimal disease at each visit, in each condition. Data was collected at weeks 2, 6 and 12.
Time Frame: Weeks 2, 6, & 12.
Population: All randomized patients were included in analyses. Missing scores within each study phase only were filled in by last observation carried forward.
Measure: Number; unit: percentage of participants
Groups:
- Corticosteroid + LCD: Corticosteroid + LCD solution applied to one side of body twice per day for 2 weeks. Then, LCD solution- only applied to one side of the body twice per day for 4 weeks.
- Corticosteroid + Placebo: Corticosteroid + placebo applied to one side of body twice per day for 2 weeks. Then, placebo-only applied to one side of the body twice per day for 4 weeks.
Arm/Group | Corticosteroid + LCD | Corticosteroid + Placebo
Number analyzed (Participants) | 15 | 15
percentage of participants
  Percentage with PGA scores ≤ 1 at Week 2 | 33.3 | 6.7
  Percentage with PGA scores ≤ 1 at Week 6 | 46.2 | 15.4
  Percentage with PGA scores ≤ 1 at Week 12 | 25.0 | 16.7

2. Secondary Outcome: Mean Percent Improvement in Disease Severity Using PGA and OTLS Scores of Target Lesions
Description: Mean percent improvement in disease severity using Physician Global Assessment (PGA) [PGA scale: Clear (0) - Very Severe (5)] and overall severity scores of target lesions (OTLS) [OTLS scale None (0) - Very Severe (4)] based on erythema, scaling and induration, at each visit interval.
Time Frame: Weeks 2, 6, & 12
Population: as for outcome 1
Measure: Mean (Full Range); unit: Mean Percent Improvement
Groups:
- Corticosteroid + LCD: Corticosteroid + LCD solution applied to one side of body twice per day for 2 weeks. Then, LCD solution-only applied to one side of the body twice per day for 4 weeks.
- Corticosteroid + Placebo: Corticosteroid + placebo solution applied to one side of body twice per day for 2 weeks. Then, placebo-only applied to one side of the body twice per day for 4 weeks.
Arm/Group | Corticosteroid + LCD | Corticosteroid + Placebo
Number analyzed (Participants) | 15 | 15
Mean Percent Improvement
  Percent improvement of PGA score at Week 2 | 39 [26 to 58] | 34 [25 to 47]
  Percent improvement of PGA score at Week 6 | 47 [34 to 72] | 25 [10 to 54]
  Percent improvement of PGA score at Week 12 | 31 [14 to 61] | 12 [-6 to 42]
  Percent improvement of OTLS score at Week 2 | 43 [31 to 59] | 43 [32 to 65]
  Percent improvement of OTLS score at Week 6 | 46 [38 to 68] | 20 [19 to 42]
  Percent improvement of OTLS score at Week 12 | 29 [14 to 56] | 7 [4 to 35]

ADVERSE EVENTS:
Time Frame: Adverse event information was monitored throughout the entire 12 week study.
Arm/Group | Corticosteroid + LCD | Corticosteroid + Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corticosteroid + LCD (N=15) | Corticosteroid + Placebo (N=15)
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — One subject was removed from the study due to a treatment-related adverse event involving contact dermatitis with clobetasol, LCD, and vehicle with bilateral itching.
Bilateral Worsening of Plaque Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Two subjects were removed from the study due to treatment-related bilateral worsening of their psoriasis.

LIMITATIONS AND CAVEATS:
This was a bilateral study in which 15 subjects total were recruited and randomized to receive both interventions simultaneously by dividing treatment arms to each side of the body.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No